CLINICAL TRIAL: NCT06409533
Title: Rate Control Efficacy in Atrial Fibrillation With Rheumatic Mitral Stenosis: Assessing Clinical Outcomes of Lenient Versus Strict Heart Rate Control in Reducing Hospitalizations, Improving Quality of Life, and Enhancing Functional Capacity
Brief Title: Rate Control Efficacy in Atrial Fibrillation With Rheumatic Mitral Stenosis: Lenient vs Strict Rate Control Strategies
Acronym: RACE-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brawijaya (Other)
Collaborators: Saiful Anwar Hospital (Other)
Responsible Party: Principal Investigator, Ardian Rizal, Ardian Rizal, MD, FIHA. Assistant Professor of Arrhythmia, Department of Cardiology and Vascular Medicine, Faculty of Medicine., University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 400/011/K.3/102.7/2023
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Rheumatic Mitral Stenosis; Arrhythmias, Cardiac
Keywords: Atrial Fibrillation; Mitral Stenosis; Rheumatic Heart Disease; Heart Rate Control; Rate Control
MeSH Terms: conditions — Atrial Fibrillation; Mitral Valve Stenosis; Arrhythmias, Cardiac; Rheumatic Heart Disease | interventions — Heart Rate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This trial implemented a double-masking protocol involving both the patients (participants) and the outcome assessors. Patients (participants) were unaware of their group assignment and the specific heart rate targets set for them. While the treating physicians (care providers) were informed about the heart rate control targets for their respective patients, the outcome assessors remained blinded to the participants' group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict Rate Control (Experimental): Physicians will aim for a resting heart rate of 60 to 80 beats per minute, as recorded by a 12-lead resting ECG after the patient has rested for 15 minutes, with the measurement taken over a one-minute period.
  Interventions: Other: Rate control
- Lenient Rate Control (Active Comparator): Physicians will aim for a resting heart rate of 81 to 110 beats per minute, as recorded by a 12-lead resting ECG after the patient has rested for 15 minutes, with the measurement taken over a one-minute period.
  Interventions: Other: Rate control

INTERVENTIONS:
Other: Rate control — Patients diagnosed with atrial fibrillation due to moderate to severe rheumatic mitral stenosis (AF-RMS) and undergoing treatment will receive care in accordance with the PERKI (Indonesian Heart Association) guidelines for Atrial Fibrillation. The selection and titration of rate control medications, including β-blockers, digoxin, or their combination, will be managed by the attending cardiologists (care providers) to achieve the target rate control.

SUMMARY:
The goal of this clinical trial is to learn if different types of heart rate control work to improve the clinical outcomes of patients with atrial fibrillation related to rheumatic mitral stenosis in terms of reducing hospitalizations, improving quality of life, and enhancing physical functional capacities. The two types of heart rate (HR) control are strict (resting HR of 60-80 bpm) versus lenient (resting HR of 81-110 bpm) rate control strategies. The main questions it aims to answer are:

* Can lenient versus strict heart rate control reduce rehospitalization in patients with atrial fibrillation and rheumatic mitral stenosis?
* Does lenient versus strict heart rate control improve the quality of life (QoL) in patients with atrial fibrillation and rheumatic mitral stenosis?
* Does lenient versus strict heart rate control enhance functional capacity in patients with atrial fibrillation and rheumatic mitral stenosis?

Researchers will compare strict rate control to lenient rate control to see if a particular rate control strategy is non-inferior to the other.

Participants will:

* Take standardized drugs as per PERKI (Indonesian Heart Association) guidelines for Atrial Fibrillation, which would be either beta-blockers, digoxin, or in combination. This standardized treatment of Atrial Fibrillation will be monitored once every month to see if the dose needs to be titrated in order to reach targeted heart rate control.
* After the target of HR control is reached, the participant will be followed up every two weeks via telephone to check for any signs and symptoms.
* Furthermore, after the HR target is reached, the participant will visit the cardiology outpatient clinics once every month for 3 consecutive months to see the clinical outcomes of hospitalization, QoL via SF-36 questionnaire, and functional capacities with 6MWT (6-minute walk test).
* Additionally, the cardiac function would be evaluated by echocardiography at the baseline (time of enrollment) and at the end of the follow up period.

DETAILED DESCRIPTION:
Rheumatic Heart Disease (RHD) often begins with untreated Group A Streptococcal infections leading to acute rheumatic fever and potentially progressing to Mitral Stenosis (MS), a condition characterized by the narrowing of the mitral valve that disrupts normal blood flow and increases atrial pressure. This pathology is closely associated with Atrial Fibrillation (AF), the most common arrhythmia in patients with MS, affecting 30-40% of such patients, with prevalence increasing with age and disease duration. The management of AF in this group focuses on anticoagulation to prevent thromboembolic events and heart rate control through medications like beta-blockers and digitalis to improve symptoms and cardiac efficiency.

Despite the guidance provided by the Rate Control Efficacy in Permanent Atrial Fibrillation (RACE II) trial, which showed non-inferiority of lenient rate control (resting heart rate <110 bpm) compared to strict control (resting heart rate <80 bpm) in reducing cardiovascular morbidity and mortality, no studies have specifically explored these strategies in patients with AF and rheumatic MS. This research gap underscores the importance of our study, aiming to assess the safety and efficacy of lenient versus strict rate control in this distinct clinical subset, potentially offering critical insights that could lead to optimized, personalized treatment protocols for these high-risk patients.

The objective of this clinical trial is to evaluate the effectiveness of different heart rate control strategies in improving clinical outcomes for patients with atrial fibrillation associated with rheumatic mitral stenosis. The outcomes of interest include reducing hospitalizations, enhancing quality of life, and improving functional capacities within three months follow-up period. The study compares two heart rate control strategies: strict control, with a target resting heart rate of 60-80 beats per minute (bpm), and lenient control, with a target resting heart rate of 81-110 bpm. The primary research questions are:

* Can lenient versus strict heart rate control reduce rehospitalization in patients with atrial fibrillation and rheumatic mitral stenosis?
* Does lenient versus strict heart rate control improve quality of life in these patients?
* Does lenient versus strict heart rate control enhance their functional capacity?

To determine whether one strategy is non-inferior to the other, researchers will compare strict and lenient rate control outcomes. Participants will:

* Receive standardized pharmacological treatment according to the PERKI (Indonesian Heart Association) guidelines for Atrial Fibrillation, potentially including beta-blockers, digoxin, or a combination thereof. This treatment regimen will be monitored monthly to adjust dosages and achieve the targeted heart rate.
* Once the target heart rate is achieved, participants will undergo bi-weekly telephone follow-ups to monitor for any signs and symptoms.
* Additionally, after reaching the heart rate target, participants will attend monthly follow-up visits at the cardiology outpatient clinic for three consecutive months to assess clinical outcomes, including hospitalization rates, quality of life via the SF-36 questionnaire, and functional capacity using the 6-minute walk test (6MWT).
* Cardiac function will be evaluated through echocardiography at the time of enrollment and at the end of the follow-up period.

The study has been approved by Health Research Ethics Committee from the main hospital (Saiful Anwar Hospital) and the satellite hospitals, i.e. Dr. Iskak Regional General Hospital and Prima Husada Sukorejo Hospital. The participants and the outcome assessors will be blinded to ensure the objectiveness, whereas the care providers would oversee the standardized treatments and heart rate control targets.

ELIGIBILITY:
Inclusion Criteria:

* Participants with atrial fibrillation and moderate-to-severe rheumatic mitral stenosis, as confirmed by ECG and echocardiography and diagnosed by the attending cardiologist.
* Patients with atrial fibrillation and severe rheumatic mitral stenosis who are ineligible for surgical intervention.
* Mean resting heart rate > 80 bpm, with or without the use of rate control medication.
* Age range between 18 and 80 years.
* Provision of informed consent by participants.

Exclusion Criteria:

* Patients with paroxysmal atrial fibrillation.
* Heart failure (HF) with unstable hemodynamics.
* HF classified as NYHA (New York Heart Association) class IV.
* Patients currently undergoing treatment for hyperthyroidism who have been euthyroid for < 3 months.
* Individuals diagnosed with a stroke, either ischemic or hemorrhagic.
* Symptomatic bradycardia accompanied by AV (atrioventricular) conduction disturbances.
* Use of a pacemaker, implantable cardioverter-defibrillator (ICD), or undergoing cardiac resynchronization therapy (CRT).
* Diagnosis of malignancy or obstructive sleep apnea (OSA).
* Patients with congenital heart defects.
* Atrial fibrillation secondary to electrolyte disturbances, hyperthyroidism, or reversible/non-cardiac causes.
* Inability to perform daily physical activities.
* Patients who have undergone CABG (coronary artery bypass graft), cardiac surgery, or a heart transplant within the past three months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Number of Hospitalizations | 0-3 months
  Patients were hospitalized at least once during the follow-up period due to worsening functional class, treated at the research hospital or at other facilities. Primary data were obtained based on the results of interviews with patients and/or their families, as well as from medical record data (numerical scale).
Quality of Life as Measured by the Short Form-36 (SF-36) Questionnaire | 3 months
  The SF-36 is a validated, patient-reported survey used widely to measure health-related quality of life. It encompasses eight scales: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The SF-36 will be measured at the end of follow up period.
Functional Capacity as Measured by 6-Minutes Walk Test (6MWT) | 3 months
  The 6MWT is a well-established, practical test widely used in clinical settings to assess the exercise tolerance and functional status of patients, particularly those with cardiovascular and pulmonary conditions. The 6MWT will be administered at the end of the study period, which is 3 months from baseline.

SECONDARY OUTCOMES:
Change of Quality of Life as Measured by the Short Form-36 (SF-36) Questionnaire | 0-3 months
  The SF-36 is a validated, patient-reported survey used widely to measure health-related quality of life. It encompasses eight scales: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health. The SF-36 will be measured twice, i.e. at the time of enrollment (baseline) and at the end of follow up period.
Change of Functional Capacity as Measured by 6-Minutes Walk Test (6MWT) | 0-3 months
  The 6MWT is a well-established, practical test widely used in clinical settings to assess the exercise tolerance and functional status of patients, particularly those with cardiovascular and pulmonary conditions. The 6MWT will be administered at baseline and at the end of the study period, which is 3 months from baseline.
Change of Metabolic Equivalents (METs) as Estimated from 6-Minutes Walk Test (6MWT) | 0-3 months
  The 6MWT measures the distance a person can walk on a flat, hard surface in a period of six minutes and is primarily used to evaluate a person's functional exercise capacity. While it is not designed to directly measure metabolic equivalents (METs), which quantify the energy cost of physical activities as a multiple of resting metabolic rate, it's possible to make a rough estimation.
  METs are a useful measure in exercise physiology because they help compare the energy expenditure of different activities. One MET is defined as the energy it costs to sit quietly, which is equivalent to a resting oxygen uptake of approximately 3.5 ml/kg/min for an average adult.
  To estimate METs, we first calculate the average speed (km/h) during the 6MWT distance (m) and use it to estimate the METs based on typical energy expenditures for walking speeds.The METs will be measured twice, i.e. at the time of enrollment (baseline) and at the end of follow up period.
Change of VO2max as Estimated from 6-Minutes Walk Test (6MWT) | 0-3 months
  Researchers have developed equations that can provide an estimated VO2max based on the distance walked during the 6MWT. These formulas take into account the fact that the distance walked in six minutes correlates with functional aerobic capacity. One such equation is:
  Estimated VO2max = (Distance in meters - 504.3)/44.73) This equation gives an estimated VO2max in mL/kg/min.
  The VO2max will be calculated at baseline and at the end of the study period, which is 3 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ardian Rizal, MD, FIHA, Principal Investigator — University of Brawijaya
Locations (3):
- Indonesia (3):
  - Saiful Anwar Hospital, Malang, East Java
  - Prima Husada Sukorejo Hospital, Pasuruan, East Java
  - Dr. Iskak Regional General Hospital, Tulungagung, East Java

IPD SHARING:
Plan to Share IPD: No
Access will be granted upon request to researchers who provide a methodologically sound proposal. The proposals should be directed to the principal investigator's office via e-mail. Approval will be contingent upon the review of the proposal and a signed data access agreement.